CLINICAL TRIAL: NCT05887557
Title: Staged Low-Barrier and Mobile Care to Improve Retention and Viral Suppression in Hard-To-Reach Vulnerable People Living With HIV
Brief Title: Multidisciplinary Low-Barrier and Mobile HIV Care to Improve Retention and Viral Suppression: Stakeholder-Engaged Design and Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: La Clínica de La Raza Inc. (Other); Lifelong Medical Care (Unknown); San Francisco AIDS Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R01AI169667 (NIH); R01AI169667 (NIH)
Record Dates: First submitted 2023-05-15; First posted 2023-06-02 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Hybrid type 2 implementation-effectiveness Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-barrier drop-in and mobile care (Other): This is a single-arm trial of a set of implementation strategies to encourage uptake of drop-in and mobile HIV care for people living with HIV who experience barriers to engage in usual scheduled appointments.
  Interventions: Other: Active Referral; Other: Drop-In Multidisciplinary HIV Care; Other: Mobile HIV Care; Other: Staged Care; Other: Identify and prepare champions at referral sites; Other: Audit and feedback at referral sites; Other: Build a coalition among referral and clinical sites; Other: Assess for readiness and identify barriers; Other: Promote adaptability; Other: Develop a formal implementation blueprint; Other: Develop educational materials; conduct ongoing training; Other: Create a learning collaborative

INTERVENTIONS:
Other: Active Referral — As an implementation science study, all clinical intervention components will be delivered as part of routine clinical care at participating clinical sites. Clinicians and staff at referral sites throughout San Francisco and Alameda counties (emergency departments, psychiatric emergency services, community clinics, care navigation and case management programs, and community-based services) will refer eligible patients who are out of care and are interested in linking to drop-in and/or mobile care services at one of the study sites. Clinical referrals will include basic patient information and contact/locator information to facilitate linkage to care. Referrals will be site-specific based on the site where the patient is interested in accessing care.
Other: Drop-In Multidisciplinary HIV Care — Each site will independently implement a drop-in multidisciplinary site-based HIV care model. Core intervention features include drop-in care (no appointments), panel management to review clinical progress for all referred patients, and case management. Each site may include adaptations to the care model determined during Aim 1 formative work.
Other: Mobile HIV Care — Each site will independently implement a mobile care model using site-specific resources. At a minimum, the mobile care team will include a clinical nurse with telemedicine (video visit) consultation with a clinician (MD/NP/PA). Mobile teams will also administer medications (including long-acting ART when available) and collect laboratory specimens (e.g. HIV viral loads)
Other: Staged Care — Clinical decision rules to escalate/de-escalate care intensity will be finalized developed during Aim 1 formative work, though will be based on a combination of clinical assessment and patient preference.
Other: Identify and prepare champions at referral sites — Identify implementation champions at each referral site. Champions will receive marketing materials to promote uptake of clinical referrals to a drop-in/mobile care site by referral site providers/staff. This strategy is aimed at improving referring provider confidence in the value of referral to the care model, reduce perceived referral complexity/improve provider capability to refer, and provide positive peer pressure to promote referrals.
Other: Audit and feedback at referral sites — Investigators will provide monthly reports to implementation champions at each referral site on aggregate number of referrals and the success of referrals (proportion linking to care). This strategy is aimed at improving perceived value of the intervention and increasing provider motivation to refer.
Other: Build a coalition among referral and clinical sites — Investigators will facilitate formation of a coalition of referral and clinic sites to improve cross-site collaboration and promote positive peer pressure to improve intra-site communication and increase referrals.
Other: Assess for readiness and identify barriers — Investigators will conduct patient in-depth interviews and clinical team focus group discussions to assess barriers to implementation of the clinical intervention. Findings from interviews and focus group discussions will inform site-specific implementation plans and adaptation of the intervention.
Other: Promote adaptability — During a co-design workshop among drop-in/mobile care site teams and site-specific meetings, the study team will collectively finalize core clinical intervention components and outline site-specific adaptations (i.e. adaptable periphery of clinical intervention).
Other: Develop a formal implementation blueprint — With each drop-in/mobile care team, develop site-specific implementation plan that includes defining care team and leadership structure, clinic workflow, implementation timeline, and progress measures. This process, and the resulting blueprint, will incorporate site-specific barriers and facilitators to implementation.
Other: Develop educational materials; conduct ongoing training — Compile a manual that includes detailed description of core intervention features, planned local adaptations, and implementation guidance. We will conduct site-specific meetings to provide training on this manual. We will also conduct regular (at least monthly) meetings between the study team and the clinic site to provide technical assistance and coaching.
Other: Create a learning collaborative — Create a cross-site learning collaborative with periodic meetings and workshops throughout the study period to facilitate cross-site communication, sharing of best practices and encourage positive peer pressure to support implementation.

SUMMARY:
The purpose of this study is to evaluate the implementation and effectiveness of a flexible, multidisciplinary, integrated drop-in/mobile HIV care approach for people living with HIV (PLH) who are not well engaged in current care systems (i.e. scheduled HIV primary care visits). The hybrid type 2 implementation-effectiveness study involves a set of implementation strategies to support implementation of the integrated drop-in/mobile HIV care approach (i.e. the evidence-informed clinical intervention) at four diverse sites in San Francisco and Alameda counties in California. Sites include an academic clinic located at a public hospital (Ward 86) and a needle exchange site (San Francisco AIDS Foundation Syringe Access Site) in San Francisco and two Federally Qualified Health Centers serving diverse patient populations in Alameda County (Trust and La Clínica). The evidence-informed clinical intervention consists of four key components: 1) active referral to care sites; 2) drop-in, multidisciplinary HIV primary care; 3) mobile HIV care; and 4) staged escalation/de-escalation of care level as needed. The study will use RE-AIM to guide evaluation, with coprimary outcomes of Reach and HIV viral suppression, and mixed methods to assess intervention Adoption, Implementation, and Maintenance. The study draws on the CFIR framework to assess site-specific implementation determinants before and after the study period. The study will undertake micro-costing using a uniform cost data collection protocol to quantify the resources needed to carry out intervention activities.

DETAILED DESCRIPTION:
Aim 1: Formative work guided by an implementation mapping process to engage key stakeholders, finalize implementation strategies to maximize successful implementation of the evidence-informed clinical intervention, and develop site specific adaptations of the interventions along with an implementation blueprint to guide intervention delivery. Proposed implementation strategies include 1) identify and prepare referral site champions, 2) audit and feedback for referral sites, 3) build a coalition between referral and study care sites, 4) assess for readiness and identify of implementation barriers at care sites, 5) adaptation of intervention components to site-specific context, 6) develop a formal implementation blueprint to guide site-specific intervention delivery, 7) develop educational materials and conduct ongoing training at each site to support implementation fidelity, and 8) create a learning collaborative to facilitate cross-site sharing of best practices and positive peer pressure.

Aim 2: Following initial formative work, a type 2 hybrid implementation-effectiveness study will be conducted using a prospective cohort of persons referred to drop-in/mobile HIV care at one of the four participating care sites (n=400). Patients are eligible for referral to the drop-in/mobile care model if they meet the following three criteria: 1) most recent HIV viral load >200 copies/mL or off ART by ≥1 month by self-report; 2) sub-optimal care engagement by self-report or chart history (defined as no current HIV primary care provider, no HIV primary care visit in the past 6 months, or ≥ 1 missed HIV primary care visit in the past 6 months); and 3) ≥1 major barrier to care engagement by self report, chart history, or clinical assessment (homelessness/unstable housing, any mental health diagnosis, any illicit substance use). The study will compare outcomes over 12 months to two propensity score-matched control groups: 1) contemporaneous patients identified using Alameda and San Francisco Departments of Public Health (DPH) HIV surveillance data (n=400) and 2) historical patients at participating clinic sites (n=400). The evaluation will be guided by the RE-AIM implementation framework, with co-primary outcomes of Reach (≥ 1 HIV primary care visit over 12 months following referral) and Effectiveness (≥1 HIV viral load <200 copies/mL over 12 months following referral).

In Aim 3: Impact Analysis to understand and model the individual, clinic, and population-level impacts of the staged care approach, the study will use several approaches: 1) Heterogeneity and Health Equity Analysis, 2) Pathway & Scenario Analysis, 3) Cost and Cost-effectiveness Analysis, and 4) Population-level Health Impact Modeling. Analyses will use mixed-methods to assess for whom the staged care approach worked and did not work and why. The Cost and Cost-effectiveness Analysis will estimate total program costs, costs associated with each intervention strategy, cost per person referred, cost per person engaged in each intervention strategy and cost per person engaged in optimized pathways. Observed study outcomes and scenario analysis results will be used to estimate the additional number of patients with suppressed viral load within the entire program, for each intervention strategy and for the identified optimized pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adults or adolescents (≥15 years) living with HIV
* Most recent HIV viral load >200 copies/mL or off ART by ≥1 month by self-report
* Sub-optimal care engagement by self-report or chart history (defined as no current HIV primary care provider, no HIV primary care visit in the past 6 months, or ≥1 missed HIV primary care visit in the past 6 months)
* ≥1 major barrier to care engagement by self report or chart history (homelessness/ unstable housing, any mental health diagnosis, any illicit substance use).

Exclusion Criteria:

Inability to give informed consent due to cognitive impairment, psychosis, or intoxication.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Reach | 12 months
  Proportion of participants who access primary HIV care over the 12 months post-referral/ propensity matching.
Number of participants with HIV viral suppression | 12 months
  Number of participants with any HIV viral load <200 copies/mL during the 12 months following referral/propensity matching.

SECONDARY OUTCOMES:
Evaluate sustained engagement in HIV care | 12 months
  Participants with ≥2 HIV primary care visits separated by ≥ 60 days with the most recent visit occurring between months 8-12.
Participants with durable viral suppression | 12 months
  Participants with ≥2 consecutive viral load measures <200 copies/mL separated by ≥60 days with most recent viral load measured during months 8-12.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Christopoulos, MD, MPH, Principal Investigator — University of California, San Francisco; Matthew Hickey, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - La Clinica de la Raza, Inc, Oakland, California
  - Lifelong Medical Care, Oakland, California
  - San Francisco AIDS Foundation, San Francisco, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified study data which includes subject demographics and study outcome measures consistent with applicable laws and regulations. Submitted data will confirm with relevant data and terminology standards and include a descriptive data dictionary of the available dataset. The primary information sharing channel for the community will be community forums, and community advisory board meetings. Prior to dissemination, all data will be fully de-identified according to standard Safe Harbor guidelines. Data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after study completion.
Access Criteria: Data will be deposited and made available through the Dryad website and these data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary data analysis study purposes.
URL: https://datadryad.org/stash

REFERENCES:
- [Derived] Garner BR, Bouris A, Charlebois ED, Li DH, Dakin A, Moskowitz J, Benbow N, Christopoulos K, Hickey MD, Imbert E. The Strategies Timeline and Activities Reporting Tables: Improving HIV Care by Improving the Reporting of Implementation Strategies. J Acquir Immune Defic Syndr. 2025 Apr 15;98(5S):e205-e215. doi: 10.1097/QAI.0000000000003613. PMID 40163072